CLINICAL TRIAL: NCT03500601
Title: Effects of Daily Tree Nut Consumption on Cognitive Function, Metabolomics and Intestinal Microbiota
Brief Title: Effects of Consumption of Nut Components on Cognitive Function, Intestinal Microbial Communities and Markers of Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: International Nut and Dried Fruit Council (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 51BQ1
Record Dates: First submitted 2018-03-12; First posted 2018-04-18 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2018-05

CONDITIONS: Cognitive Function; Urinary Metabolites; Intestinal Microbiota
Keywords: Cognition; Metagenomics; Metabolomics

STUDY DESIGN:
Intervention Model Description: 2 x 4 week intervention with 4 week washout
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): Nut components
  Interventions: Other: Nut components
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Nut components — nut components consumed daily for a period of 28 days
  Arms: Active treatment
Other: Placebo — Placebo consumed daily for a period of 28 days
  Arms: Placebo

SUMMARY:
Tree nuts (for example brazil nuts, almonds, hazelnuts, walnuts, cashew nuts etc) contain a wide variety of nutrients including fatty acids, polyphenols and micronutrients. The beneficial health effects ascribed to the consumption of tree nuts include improvements to cardiovascular outcomes and regulation of glucose levels and inflammation. Emerging evidence suggests that specific components of nuts may also contribute to brain health and function.

The aim of the present study is to assess the effects of four weeks' supplementation of nut components on cognition and subjective measures. Urinary metabolites and intestinal microbial communities will also be assessed allowing biomarkers of nut exposure to be highlighted.

DETAILED DESCRIPTION:
To date, only two small human intervention trials have evaluated the effects of nuts as a sole intervention on cognition. One study reported a benefit verbal fluency and constructional praxis following daily consumption of 6 g brazil nuts for 6 months in older adults diagnosed with mild cognitive impairment. Eight weeks' consumption of 60 g/d walnuts in healthy young adults aged 18-25 years also resulted in improved inferential verbal reasoning scores compared to placebo.

The development of various 'omics' technologies has enabled researchers to investigate the influence of nutrients or dietary change on metabolic pathways at multiple levels with a view to developing biological markers of dietary intake.

Metabolomic approaches have been used successfully to study nut consumption; for example putative biomarkers of nut consumption have been revealed as metabolites associated with serotonin pathways. Furthermore, certain nut biomarkers identified using metabolomics appear to be negatively associated with health parameters which is suggested to be due to gut microbiota dysbiosis and provides an important link between nut consumption, the gut microflora and metabolic pathways.

This study will assess the effects of four weeks' supplementation with nut components on cognition. Metabolomic and metagenomic approaches will be utilised to analyse urinary metabolites and intestinal microbial communities allowing biomarkers of nut exposure to be highlighted. Metabolic and gut microbiota responses will then be correlated with changes in cognition in order to identify inter-individual differences in response, and further understanding of the mechanisms underpinning cognitive benefits of nut consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Willing to abstain throughout the trial from any nutritional supplementation
* Willing to abstain throughout the trial from the intake of any nuts or nut containing products

Exclusion Criteria:

* Aged under 18 or over 49
* Relevant pre-existing medical condition/illness
* Current use of prescription medications (excluding contraception)
* Learning difficulties and dyslexia
* Visual impairment that cannot be corrected with glasses or contact lenses including colour blindness
* Currently suffer from migraines (> 1 per month)
* Smoking or use of any nicotine replacement products e.g. vaping, gum, patches
* History of or any current food intolerances/sensitivities, including nut/peanut allergies
* Never consumed nuts, or regularly consume nuts more than twice per week
* Irregular bowel function (less than one bowel movement per day)
* Body mass index (BMI) under 18.5 or over 30
* Pregnancy, seeking to become pregnant, or current lactation
* Inability to complete all of the study assessments
* Current participation in other clinical or nutrition intervention studies
* Not proficient in English equivalent to IELTS band 6 or above
* Have any known active infections
* Blood pressure >139/89mmHg
* Are employed in a job that includes night shift work
* Have habitually used supplements within the last month (defined as more than 3 consecutive days or 4 days in total)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Logical reasoning | At 28 days post dose, adjusted for baseline
  Cognition - executive function

SECONDARY OUTCOMES:
Location learning | At 28 days post dose, adjusted for baseline
  Cognition - spatial memory
Choice reaction time | At 28 days post dose, adjusted for baseline
  Cognition - attention
Rapid Visual Information Processing | At 28 days post dose, adjusted for baseline
  Cognition - working memory
Numeric working memory | At 28 days post dose, adjusted for baseline
  Cognition - working memory
Stroop | At 28 days post dose, adjusted for baseline
  Cognition - executive function
Peg and Ball | At 28 days post dose, adjusted for baseline
  Cognition - executive function
Word recall | At 28 days post dose, adjusted for baseline
  Cognition - episodic memory
Word recognition | At 28 days post dose, adjusted for baseline
  Cognition - episodic memory
Picture recognition | At 28 days post dose, adjusted for baseline
  Cognition - episodic memory
Bond-Lader | At 28 days post dose, adjusted for baseline
  Mood
Profile of Mood States (POMS) | At 28 days post dose, adjusted for baseline
  Mood
Urinary metabolites (fingerprinting and profiling) | At 28 days post dose, adjusted for baseline
  Liquid chromatography/mass spectrometry, combined with data mining using specific software to identify specific metabolites influenced by supplementation
Intestinal microbial communities | At 28 days post dose, adjusted for baseline
  Analysis of total DNA using standardised procedures targeting bacteria using the 16S rRNA gene.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Haskell-Ramsay, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne & Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rita Cardoso B, Apolinario D, da Silva Bandeira V, Busse AL, Magaldi RM, Jacob-Filho W, Cozzolino SM. Effects of Brazil nut consumption on selenium status and cognitive performance in older adults with mild cognitive impairment: a randomized controlled pilot trial. Eur J Nutr. 2016 Feb;55(1):107-16. doi: 10.1007/s00394-014-0829-2. Epub 2015 Jan 8. PMID 25567069
- [Background] Pribis P, Bailey RN, Russell AA, Kilsby MA, Hernandez M, Craig WJ, Grajales T, Shavlik DJ, Sabate J. Effects of walnut consumption on cognitive performance in young adults. Br J Nutr. 2012 May;107(9):1393-401. doi: 10.1017/S0007114511004302. Epub 2011 Sep 19. PMID 21923981
- [Background] Tulipani S, Llorach R, Jauregui O, Lopez-Uriarte P, Garcia-Aloy M, Bullo M, Salas-Salvado J, Andres-Lacueva C. Metabolomics unveils urinary changes in subjects with metabolic syndrome following 12-week nut consumption. J Proteome Res. 2011 Nov 4;10(11):5047-58. doi: 10.1021/pr200514h. Epub 2011 Sep 29. PMID 21905751
- [Background] Mora-Cubillos X, Tulipani S, Garcia-Aloy M, Bullo M, Tinahones FJ, Andres-Lacueva C. Plasma metabolomic biomarkers of mixed nuts exposure inversely correlate with severity of metabolic syndrome. Mol Nutr Food Res. 2015 Dec;59(12):2480-90. doi: 10.1002/mnfr.201500549. Epub 2015 Oct 21. PMID 26412215
- [Derived] Haskell-Ramsay CF, Dodd FL, Smith D, Cuthbertson L, Nelson A, Lodge JK, Jackson PA. Mixed Tree Nuts, Cognition, and Gut Microbiota: A 4-Week, Placebo-Controlled, Randomized Crossover Trial in Healthy Nonelderly Adults. J Nutr. 2023 Jan 14;152(12):2778-2788. doi: 10.1093/jn/nxac228. PMID 36202391